CLINICAL TRIAL: NCT07407738
Title: ShockFast Intravascular Lithotripsy Device for Treatment of Calcified Coronary Lesions, a Prospective, Randomised, International Trial: ShockFast IVL Trial
Brief Title: ShockFast Intravascular Lithotripsy Device for Treatment of Calcified Coronary Lesions
Acronym: IVL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shunmei Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3W RCG 1
Record Dates: First submitted 2026-01-29; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Coronary Arterial Disease; Calcified Coronary Artery Disease
Keywords: Shockwave Intravascular Lithotripsy; Shockfast Intravascular Lithotripsy; Coronary Calcified Lesion; IVL

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shockfast IVL (Experimental): Interventional procedure using a dedicated device to treat coronary calcified lesions by offering precise control of sonic pressure waves for safe fracture calcium deposits within the artery walls, thus maintaining vessel flexibility and promoting smoother stent placement. The ShockFast device has an improved crossing profile and 2 lengths of the catheter: 12 and also 15mm compared to ShockWave which has only 1 length.
  Interventions: Device: Shockfast IVL
- Shockwave IVL (Active Comparator): Interventional procedure that utilizes a fluid-filled catheter connected to an energy source that generates mechanistically tuned ultrasonic acoustic pressure waves - or Shockwaves - for modification, fracture, and fragmentation of vascular calcification.
  Interventions: Device: Shockwave IVL

INTERVENTIONS:
Device: Shockwave IVL — Treatment of subjects with coronary calcified lesions with an interventional procedure that utilizes a fluid-filled catheter connected to an energy source that generates mechanistically tuned ultrasonic acoustic pressure waves - or Shockwaves - for modification, fracture, and fragmentation of vascular calcification.
  Arms: Shockwave IVL
Device: Shockfast IVL — Treatment of subjects with coronary calcified lesions with an interventional procedure using a dedicated device to treat coronary calcified lesions by offering precise control of sonic pressure waves for safe fracture calcium deposits within the artery walls, thus maintaining vessel flexibility and promoting smoother stent placement. The ShockFast device has an improved crossing profile and 2 lengths of the catheter: 12 and also 15mm compared to ShockWave which has only 1 length.
  Arms: Shockfast IVL

SUMMARY:
Coronary artery disease is caused by narrowing of the artery lumen. Treatment with Percutaneous Coronary Intervention (PCI) may be needed. This is a minimally invasive procedure used to treat narrowed or blocked coronary arteries. Sometimes a stent is placed to keep the artery open. If the lesions in the coronary artery are calcified, this may cause difficulties for successful stent placement. The calcified plaques can be fractured via intravascular lithotripsy (IVL) with devices like ShockWave IVL and ShockFast IVL. The aim of this study is to compare the this relatively new ShockFast IVl with the more widely used ShockWave IVL.

DETAILED DESCRIPTION:
Coronary calcified lesions have evolved as one of the most challenging indications for coronary percutaneous interventions (PCI). Different dedicated devices have been recently introduced into the market to improve procedural success in this challenging PCI population. Shockwave Intravascular Lithotripsy, (Shockwave IVL), Shockwave Medical, SC, CA, USA, was the first intracoronary device that used sonic pressure to fracture intracoronary calcium. The device safety and efficacy has been proved in a series of clinical trials. ShockFast intravascular lithotripsy (ShockFast IVL), Shunmei medical, Shenzhen, China, is a new dedicated device to treat intracoronary calcium that makes use of sonic pressure waves to fracture calcified plaques. ShockFast IVL has recently obtained CE mark approval for this indication.

The aim of this study is to compare this new lithotripsy device (ShockFast IVL) with the existing and widely used lithotripsy device that uses the same principle of action, the Shockwave IVL, Shockwave Medical, SC, CA, USA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years undergoing PCI for stable or unstable angina or staged procedure after successful treatment of a myocardial infarction where heart enzymes are decreasing

   Angiographic criteria:
2. Native de novo coronary lesions
3. Vessel diameter between 2.5mm - 4.0mm
4. Lesion Length: ≤40mm
5. Severe Calcification:

   1. Calcification visible on the upper and the lower sides of the vessel wall in at least two angiographic projections that differ ≥ 60° from each other
   2. Presence of severe calcified protruding noduli
6. No flow disturbances at baseline (Thrombolysis in Myocardial Infarction [TIMI] 3 flow at baseline)
7. Target lesion with diameter stenosis ≥70% by visual, or ≥50% with evidence of clinical ischemia

   OCT Criteria:
8. Total calcium arc > 180° or
9. Presence of a protruding calcified noduli

Exclusion Criteria:

1. Ejection fraction less than 25%
2. Lesion located in Left Main (LM) coronary artery
3. Calcifications located mostly > 0.5 mm from the vessel lumen.
4. Severe renal Impairment; Serum Creatinine > 220 μmol or currently undergoing hemodialysis
5. Severe lesion tortuosity where OCT is judged impossible to cross.
6. Inability to tolerate dual antiplatelet therapy for 6 months or longer
7. Inability to obtain inform consent or deemed poorly compliant by the investigator
8. Presence of permanent pacemaker
9. Angiographic evidence of thrombus in the target vessel
10. Target lesion located at or involving within 5mm of the coronary ostium of the Left Anterior Descending artery (LAD), Left Circumflex artery (LCX)
11. Target lesion is a chronic total occlusion (CTO)
12. Presence of aneurysm within 10mm proximal or distal to the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Stent area post PCI measured at the minimal lumen area during initial procedure, evaluated by OCT | Hospitalisation (during procedure)

SECONDARY OUTCOMES:
Target lesion failure defined as cardiac death, target-vessel myocardial infarction and target-lesion revascularisation at discharge and 30 days | 30 day follow-up
Angiographic success | Hospitalisation (during procedure)
  * Defined as a successful stent delivery with diameter of stenosis post PCI of <50% without severe dissection (type D-F), perforation, abrupt vessel closure or persistent less than Thrombolysis in Myocardial Infarction (TIMI)-3 flow.
  * By collecting data through angiography and imaging:
    * Minimal lumen area post stenting
    * Residual area of stenosis
    * Residual diameter of stenosis <30%
    * Residual diameter of stenosis <50%
    * Optical Coherence Tomography (OCT) measured under expansion (<80% of the reference lumen area)
    * Post-IVL acute area gain (measured at the minimum lumen area post IVL)
    * Number of visible calcium cracks post IVL
    * Severe coronary dissection post IVL (type C-F)
Device success | Hospitalisation (during procedure)
  Defined as success of the device to cross and fully expand

CONTACTS AND LOCATIONS:
Locations (11):
- France (3):
  - Infirmerie Protestante de Lyon, Lyon
  - Centre Cardiologique du Nord, Paris
  - Centre Hospitalier de Valenciennes, Valenciennes
- Poland (4):
  - Medical University of Silesia, Katowice
  - University Hospital Krakow, Krakow
  - Miedziowe Centrum Zdrowia, Lubin
  - Regional Specialist Hospital, Wroclaw
- Spain (4):
  - La Paz University Hospital, Madrid
  - La Princesa Univeristy Hospital, Madrid
  - Virgen Arrixaca University Clinical Hospital, Murcia
  - Virgen del Rocío University Hospital, Seville

IPD SHARING:
Plan to Share IPD: No